CLINICAL TRIAL: NCT01954927
Title: Pain Management of Vaso-Occlusive Crisis in Children and Young Adults With Sickle Cell Disease
Brief Title: Pain Management in Children and Young Adults With Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Scan | Design Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMVOC
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2018-07

CONDITIONS: Sickle Cell Disease
Keywords: Pain control
MeSH Terms: conditions — Anemia, Sickle Cell; Agnosia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Active Comparator): Patients will be randomized to receive one dose of gabapentin.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Patients will be randomized to receive one dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin is supplied as an oral suspension. Patients randomized to the gabapentin arm will receive a single dose of gabapentin as soon after enrollment as feasible. The gabapentin dose will be given orally and will be approximately 15 mg/kg with a maximum dose of 900 mg.
  Other Names: Neurontin(R)
  Arms: Gabapentin
Drug: Placebo — Placebo will be prepared by the SJCRH pharmacy and will be similar in appearance, quantity and taste to the gabapentin drug. Patients randomized to the placebo arm will receive a single dose of placebo as soon after enrollment as feasible. The placebo dose will be given orally and will be approximately 15 mg/kg with a maximum dose of 900mg.
  Arms: Placebo

SUMMARY:
This is a phase II double-blind placebo-controlled clinical trial evaluating the effect of gabapentin when added to standard pain management for patients with sickle cell disease experiencing acute pain crisis in the ambulatory care setting.

Sickle cell pain is different for every patient. Some patients get complete relief from routine pain medicines, and others need more time or more doses of pain medicines before the pain goes away completely. It is known that humans have many types of pain, including something called neuropathic pain. Neuropathic pain in other conditions (such as diabetes) has been treated successfully with a medicine called gabapentin. The investigators in this study suspect that some sickle cell pain is a combination of pain types. They would like to see if adding gabapentin to the usual pain medicines makes pain go away faster or more completely.

Primary Objective:

* To assess the analgesic efficacy of gabapentin vs. placebo for pain during vaso-occlusive crisis (VOC) in participants with sickle cell disease (SCD). A response to study drug will be defined by a decrease in pain score of ≥ 33% between presentation to the acute care setting and assessment at 3 hours post administration of study drug.

Secondary Objective:

* To compare the total morphine equivalent dose (mg/kg) used to control pain during VOC between presentation to the acute care setting and assessment at 3 hours post administration of study drug in the gabapentin vs. placebo groups.

DETAILED DESCRIPTION:
Upon participant enrollment, study staff will randomize the participant to one of 2 possible treatment arms: a single dose of gabapentin or a single dose of placebo. Morphine or other opioid and non-steroidal anti-inflammatory drugs will be available to both groups as needed for pain and will be administered according to the current standard of care for pain in VOC from the Department of Hematology at St. Jude Children's Research Hospital (SJCRH). Randomization will be performed in the SJCRH pharmacy by a pharmacist. The randomization will be stratified by three age categories (1-3 years of age, 4-6 years, and 7 years or older) for which distinct pain assessment tools are applied and for 2 pain score categories at assessment at presentation (4-6 and 7-10, respectively). A block randomization with block sizes varying randomly between 4 and 6 will be used in each stratum.

Pain scores will be obtained at presentation to the acute care setting and 3 hours (± 15 minutes) post administration of study drug. Participants who were discharged will be contacted by study staff between 24 and 72 hours following administration of study drug to see if there have been any side effects. Patients who were admitted after administration of the study drug will be monitored through hospital record to determine if any unexpected events occurred. After this follow up, participation in the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have sickle cell disease (any genotype) documented in the St. Jude medical record.
* Participant must be seeking care for acute vaso-occlusive pain at St. Jude Children's Research Hospital.
* Participant age must be ≥1 year and <21 years.

Exclusion Criteria:

* Prior randomization in this study.
* Mild pain (score <4) or pain for which treatment with opioid is not indicated.
* Pregnant or lactating female.
* Decreased glomerular filtration rate (GFT) (<60ml/min/1.73m^2) as estimated by the revised Schwartz equation.
* Current treatment with gabapentinoid drugs (gabapentin or pregabalin).
* Known seizure disorder.
* Current treatment with antiepileptic agents.
* Pain in combination with other clinical symptoms that require additional interventions, including fever with focus, acute chest syndrome, acute injury, or splenic sequestration.
* Allergy to gabapentin.
* Current participation in another research study with an investigational new drug/device (IND/IDE) agent.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doralina Anghelescu, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants meeting eligibility criteria were enrolled between 10/7/2013 to 1/3/2018. They were randomized to either gabapentin or placebo.
Pre-assignment Details: The study was stopped early due to slow accrual when there were 82 patients with evaluable pain assessments available for the primary objective. Patients asleep at pain assessment times led to missing pain assessments.
Groups:
- Gabapentin: Participants were randomized to receive one dose of gabapentin.
  Gabapentin: Gabapentin is supplied as an oral suspension. Patients randomized to the gabapentin arm received a single dose of gabapentin as soon after enrollment as feasible, given orally, approximately 15 milligram/kilogram (mg/kg) with a maximum dose of 900 milligram (mg).
- Placebo: Participants were randomized to receive one dose of placebo.
  Placebo: Placebo was prepared by the SJCRH pharmacy, similar in appearance, quantity and taste to the gabapentin drug. Patients randomized to the placebo arm received a single dose of placebo as soon after enrollment as feasible, given orally, in a volume that matched the active medication arm.
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 45 | 45
Completed | 42 | 44
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 42 | 81
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11.9 [8.2 to 15.6] | 14.3 [7.7 to 16.3] | 12.4 [8.1 to 15.8]
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (4.5) | 11.8 (5.3) | 11.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 22 | 35
  Male | 29 | 22 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 42 | 44 | 86
  Non-Spanish speaking Non Hispanic | 40 | 44 | 84
  Unknown | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 42 | 44 | 86
Sickle cell genotype [Count of Participants; unit: Participants]
  SBeta Zero Thalassemia | 6 | 2 | 8
  Hemoglobin SC | 10 | 15 | 25
  Hemoglobin SS | 18 | 26 | 44
  Other | 8 | 1 | 9
Pain score category at presentation [Count of Participants; unit: Participants] — (0=no pain and 10=worst possible pain)
  Participants
    4-6 | 10 | 12 | 22
    7-10 | 32 | 32 | 64
Pain at presentation (before randomization) [Mean (Standard Deviation); unit: units on a scale] — (0=no pain and 10=worst possible pain)
  units on a scale | 8.0 (1.6) | 7.7 (1.9) | 7.8 (1.8)
Pain at presentation (before randomization) [Median (Inter-Quartile Range); unit: units on a scale] — (0=no pain and 10=worst possible pain)
  units on a scale | 8.0 [7.0 to 10.0] | 8.0 [6.5 to 10.0] | 8.0 [7.0 to 10.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Pain Interventions by Arm Between Presentation and 3 Hours Post Administration of Study Drug
Description: Pain scales used are the numerical rating system, the Faces Pain Scale, and the Faces, Legs, Arms, Cry and Consolability (FLACC) pain scale (for patients 7 years or older, ages 4-6 years, or less than 4 years, respectively). For each patient, if the reduction of the pain scores (0=no pain and 10=worst possible pain) between presentation to the acute care setting and 3 hours post administration of study drug is 33% or greater, then this patient will be defined as having a successful intervention. The proportions of successful interventions in the gabapentin and placebo groups will be estimated and compared using Z-test.
Time Frame: Baseline and 3 hours (±30 minutes) post administration of study drug. The 3-hour pain assessment time-period was extended for subjects that were sleep until the first available measurement.
Population: Patients with Sickle cell disease (any genotype) ages ≥1 year and <21 years seeking care for acute vaso-occlusive pain at St Jude Children's Hospital. A total of 4 subjects were missing the pain assessment at 3 hours (2 in each arm). The resulting sample sizes were n=40 (Gabapentin arm) and n=42 (placebo arm), for a total sample size of n=82.
Measure: Count of Participants; unit: Participants
Groups:
- Gabapentin: Participants were randomized to receive one dose of gabapentin.
  Gabapentin: Gabapentin is supplied as an oral suspension. Patients randomized to the gabapentin arm received a single dose of gabapentin as soon after enrollment as feasible, given orally, approximately 15 mg/kg with a maximum dose of 900 mg.
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 40 | 42
Participants
  No | 13 | 17
  Yes | 27 | 25
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.227, z-test Proportion — 1-sided p-value; z-test of proportions without continuity correction

2. Secondary Outcome: Morphine Equivalent Doses Administered From Presentation to 3-hours Post Treatment With Gabapentin/Placebo
Description: The equivalent dose of morphine in mg
Time Frame: The 3-hour pain assessment was the pain assessment closest in time to the 3-hour time and was typically within 30 minutes of target. The time period was extended for 12 patients that were sleeping.
Population: Patients with Sickle cell disease (any genotype) ages ≥1 year and <21 years seeking care for acute vaso-occlusive pain at St Jude Children's Hospital.
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 44
mg/kg | 0.12 [0.09 to 0.22] | 0.13 [0.09 to 0.22]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.897, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Number of Participants With Successful Pain Interventions by Arm Between Presentation and Point of Decision for Either Hospital Admission or Discharge to Home
Description: For each patient, if the reduction of the pain scores (0=no pain and 10=worst possible pain) between presentation to the acute care setting and Point of decision for either hospital admission or discharge to home is 33% or greater, then this patient will be defined as having a successful intervention.
Time Frame: From time of presentation to the acute care setting until time of either discharge to home or admission to the hospital, up to 8 hours.
Population: Patients with Sickle cell disease (any genotype) ages ≥1 year and <21 years seeking care for acute vaso-occlusive pain at St Jude Children's Hospital. There were 2 subjects in the Gabapentin group that did not have a pain assessment admit/discharge decision. N=84 patients had assessments at both presentation and admit/discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 40 | 44
Participants
  No | 10 | 17
  Yes | 30 | 27
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.181, Chi-squared

4. Other Pre Specified Outcome: Morphine Equivalent Doses Administered From Presentation to the Point of Decision for Either Admission or Discharge to Home
Description: To compare the total morphine equivalent dose (mg/kg) used to control pain during VOC between presentation to the acute care setting and the point of decision for either admission or discharge to home, in the gabapentin and placebo groups.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 44
mg/kg | 0.13 [0.10 to 0.25] | 0.13 [0.09 to 0.25]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.730, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Hospital Admission
Description: To compare the rate of admission related to pain management, in the gabapentin vs. placebo groups. (Outcome: binary response - admitted or discharged)
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 44
Participants
  No | 32 | 32
  Yes | 10 | 12
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.713, Chi-squared

6. Other Pre Specified Outcome: Absolute Change in Pain From Study Drug to 3 Hours Post Administration of Study Drug
Description: To compare the change in pain score from time of administration of study drug to assessment at 3 hours post administration of study drug in the gabapentin vs. placebo groups. (0=no pain and 10=worst possible pain)
Time Frame: Study drug administration to 3-hours post study drug administration
Population: Patients with Sickle cell disease (any genotype) ages ≥1 year and <21 years seeking care for acute vaso-occlusive pain at St Jude Children's Hospital. Placebo arm: 6 subjects missed pain assessments at treatment; 2 missed pain assessment at 3h. Gabapentin arm: 7 missed pain assessment at treatment; 2 of the 7 also missed the assessment at 3h.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 35 | 36
score on a scale | 0 [0 to 2] | 0.5 [0 to 2]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.739, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Absolute Change in Pain, Study Drug to Hospital Discharge Decision
Description: To compare the change in pain score from time of administration of study drug to the point of decision for either admission or discharge to home, in the gabapentin and placebo groups. (0=no pain and 10=worst possible pain)
Time Frame: as for outcome 3
Population: Patients with Sickle cell disease (any genotype) ages ≥1 year and <21 years seeking care for acute vaso-occlusive pain at St Jude Children's Hospital. Placebo arm: 6 subjects missed pain assessments at treatment. Gabapentin arm: 7 subjects missed pain assessment at treatment; 2 of the 7 missed the assessment at hospital discharge decision.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 35 | 38
score on a scale | 1.0 [0.0 to 3.0] | 0.5 [0.0 to 2.0]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.388, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated by one phone contact within the following 72 hours.
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 5/42 | 2/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=42) | Placebo (N=44)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT01954927/Prot_SAP_000.pdf